CLINICAL TRIAL: NCT00211913
Title: A Multicenter, Randomized, Placebo-Controlled, Double-Blinded Study to Evaluate Safety and Immunogenicity of StaphVAX®, a Bivalent Staphylococcus Aureus Glycoconjugate Vaccine, in Adult Patients Undergoing Cardiovascular Surgery
Brief Title: StaphVAX in Cardiovascular Surgery Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nabi Biopharmaceuticals (Industry)
Responsible Party: Matt Hohenboken, MD, PhD, Executive Director Clinical & Medical Affairs, Nai Biopharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Nabi-1366
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2008-01-04 (Estimated); Status verified 2007-12

CONDITIONS: Staphylococcal Infections; Cardiovascular Diseases; Cardiovascular Surgical Procedures
MeSH Terms: conditions — Staphylococcal Infections; Cardiovascular Diseases | interventions — StaphVax

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- vaccine (Experimental): single dose of StaphVAX®
  Interventions: Biological: S. aureus Type 5 & 8 Capsular Polysaccharide Conjugate
- placebo (Placebo Comparator): single dose
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: S. aureus Type 5 & 8 Capsular Polysaccharide Conjugate — single IM dose totalling 200 mcg of conjugate
  Other Names: StaphVAX®
  Arms: vaccine
Biological: placebo — single IM dose
  Arms: placebo

SUMMARY:
S. aureus is the most common pathogen encountered in infection associated with cardiovascular surgery. StaphVAX® is a bivalent S. aureus types 5 and 8 vaccine which contains the purified capsular polysaccharides (CPS) that have been implicated as a major factor in the invasiveness of S. aureus. Immunoprophylaxis by vaccinating against S. aureus prior to surgery could provide sufficient antibody concentrations during surgery and during the wound healing period so as to decrease the risk of S. aureus infection. This study aims to demonstrate the immunogenicity and safety of a single dose of StaphVAX in patients who are candidates for cardiovascular surgery.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for cardiovascular surgery
* Expected to comply with protocol
* Negative pregnancy test where appropriate
* Written informed consent

Exclusion Criteria:

* Known S. aureus infection in past 3 months
* Known infection in the past 2 weeks
* Known HIV infection
* Pregnancy or breast-feeding
* Immunomodulatory drugs
* Malignancy or treatment for malignancy within the past six months, other than basal cell, localized squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or early stage prostate cancer
* investigational drugs, vaccines or products in the past 30 days
* Hypersensitivity to components of StaphVAX

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2004-06; Primary Completion 2005-10 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Serotype-specific antibody concentrations | 6 weeks after the vaccine dose

SECONDARY OUTCOMES:
Serotype-specific antibody concentrations | at other time points 7-180 days after the vaccine dose.
adverse events | 0-180 days after vaccine dose

CONTACTS AND LOCATIONS:
Overall Officials: Preston Holley, MD, Study Director — Nabi Biopharmaceuticals
Locations (1):
- Clinical Research Associates of Tidewater, Norfolk, Virginia, United States